CLINICAL TRIAL: NCT01356485
Title: A Multi-center, Randomized, Double Blind, Dose Escalation Safety Study of MP4CO in Clinically Stable Adult Sickle Cell Patients
Brief Title: Safety Study of MP4CO in Adult Sickle Cell Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sangart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: SCD-105
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Anemia, Sickle Cell; Sickle Cell Anemia; Sickle Cell Disease; Sickle Cell Disorders; Hemoglobin SC Disease; Sickle Cell Hemoglobin C Disease
Keywords: Sickle cell anemia; Sickle cell disease; Sickling crisis; Vaso-occlusive crisis; Carboxyhemoglobin; Oxygen therapeutic; Hemoglobin solutions; Pegylated hemoglobin
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease; Vaso-Occlusive Crises | interventions — PEGylated carboxyhemoglobin bovine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MP4CO (Experimental): Escalating doses of MP4CO, administered intravenously
  Interventions: Drug: MP4CO
- Saline (Placebo Comparator): Normal saline (0.9% sodium chloride solution)
  Interventions: Drug: Sodium chloride solution

INTERVENTIONS:
Drug: MP4CO — 43 mg/mL pegylated carboxyhemoglobin [≥ 90% CO hemoglobin saturation] in physiological acetate electrolyte solution
  Other Names: Pegylated carboxyhemoglobin; PEG carboxyhemoglobin
  Arms: MP4CO
Drug: Sodium chloride solution — Normal saline (0.9% sodium chloride solution)
  Other Names: Normal saline; Sodium chloride; 0.9% NaCL solution
  Arms: Saline

SUMMARY:
Sickle Cell Anemia is caused by an inherited hemoglobin disorder. Healthy red blood cells are discoid and can deform and move through small blood vessels to carry oxygen to all parts of the body. In sickle cell disease, as red blood cells circulate and oxygen is released in the circulatory system, the deoxygenated abnormal hemoglobin S can begin to polymerize. When this occurs, the red blood cells can become sticky and elongated. These sickled red blood cells are less flexible and will obstruct small blood vessels and block normal red blood cells from traveling through the circulatory system, which limits oxygen delivery to tissues and organs. This is known as a "sickle crisis".

Patients suffering from a sickle crisis experience severe pain and are at risk of stroke, heart attack or even death. By lowering the level of oxygen pressure at which sickling occurs and opening the vasculature and rapidly delivering oxygen directly to ischemic tissues, the addition of MP4CO to existing treatment protocols may alleviate pain associated with a sickle cell crisis, abort a crisis and/or potentially reduce the duration of a crisis. This could mean less time in the hospital and an improved quality of life for patients with sickle cell anemia.

DETAILED DESCRIPTION:
To date, no specific agent has been approved to treat sickle cell crisis, to reduce the severity of a sickling crisis, or to shorten the duration of admission. Current therapy for a sickling crisis is limited to hydration and symptomatic pain relief with opiates when pain is severe enough to cause admission to hospital. Administration of oxygen by inhalation alone has not proven effective. Carbon monoxide (CO) binds to Hb S and, while attached, prevents and reverses polymerization of Hb S chains and consequent distortion of the red blood cell. Carbon monoxide at very low doses also acts as a messenger to cells, reducing inflammation, reducing oxygen requirements, and preventing programmed cell death (apoptosis).

The MP4 molecule can be modified to carry CO and other gases to enhance therapeutic benefit for certain patients. MP4CO is therefore designed to deliver therapeutic, non-toxic levels of CO, to provide an immediate metabolic signal to cells and to reduce inflammation. Once the CO is released from the compound, the MP4 molecule gets oxygenated in the lung and then delivers oxygen to ischemic tissues.

Previously published studies provide a good foundation to postulate that a chemically modified hemoglobin such as MP4CO might have the ideal properties as an oxygen therapeutic agent for treatment or reversal of a sickling crisis. The initial release of CO from MP4CO is predicted to have a therapeutic effect including immediate stabilization of Hb S to prevent further polymerization and reverse existing sickling, vasodilation of capillaries, and anti-inflammatory properties. The subsequent circulation of the MP4 molecule as an oxygen therapeutic agent (after converting to MP4OX following oxygenation in the lungs) will help to 1) preferentially oxygenate ischemic cells, 2) reverse partially sickled red cells, and 3) improve oxygenation of local tissues, thereby potentially ameliorating the painful VOC caused by red blood cell sickling. In addition, MP4CO has enhanced chemical stability, which enables storage at room temperature while minimizing methemoglobin formation.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients (18 years of age or older) with diagnosed sickle cell disease based on Hb SS, or S/β0 Thalassemia genotype, who are clinically stable and not experiencing an acute episode of pain

Exclusion Criteria:

* At least 4 painful VOCs within the preceding year requiring hospital treatment
* Urgent care facility, hospital treatment or admission for treatment of a painful VOC within the previous 2 months
* History of a painful VOC lasting longer than 2 weeks or > 12 pain episodes requiring intervention in a medical facility (emergency room, urgent care or clinic) in preceding year
* Baseline VAS pain score ≥ 4 cm
* Hemoglobin < 6 g/dL
* Transfusion of packed red blood cells within previous 4 weeks
* Currently on iron chelation therapy
* History of sickle cell disease-attributed CNS disease (including a) recent or past history of stroke; b) ongoing treatment with chronic transfusion therapy to prevent stroke; c. history of seizures or epilepsy; and d. evidence of or known overt cerebral vasculopathy or known cerebral vessel narrowing
* Evidence of pulmonary hypertension, based on an estimated systolic pulmonary artery pressure > 25 mmHg calculated from TRJ velocity from a transthoracic echocardiography (TTE) assessment at Screening visit or from a previous TTE assessment if it was done within 1 year prior to randomization
* Baseline oxygen saturation by pulse oximetry ≤ 90%
* History of a priapism within the last year
* History of hypertension requiring anti-hypertensive therapy
* Baseline bradycardia (heart rate < 60/min)
* History of myocardial infarction, myocardial ischemia, or angina
* Renal dysfunction or creatinine level within past 6 weeks of ≥ 1.2 mg/dL (≥ 106 µmol/L) or a urine protein/creatinine ratio (PCR) > 50 mg/mmol
* Hepatic dysfunction (AST or GGT > 3x ULN, or ALT >2x ULN, or conjugated bilirubin > 2x patient's baseline within the last 6 weeks)
* Positive pregnancy test
* Any acute or chronic condition which would limit the patient's ability to complete the study
* Evidence of, or known to be chronically abusing illegal drugs or excessive quantities of alcohol
* Known to have HIV, or active Hepatitis B or C infection, or tuberculosis
* Received any other investigational drug(s) within 30 days prior to randomization
* Professional or ancillary personnel involved with this study or in the employment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
No efficacy evaluations will be made in this safety study | 28 days

SECONDARY OUTCOMES:
Adverse events | From 0 hrs after dosing through 28 Day Follow-up visit
Vital signs | Baseline, Hourly from 0 - 8 hours, 24, 48, and 72 hours, and at 7 days
  Blood pressure, heart rate, respiration, temperature
Laboratory assessments | Baseline, 24, 48, and 72 hours, and at 7 days
  Hematology, serum chemistry, urinalysis, renal function and biomarkers
Pain levels | Baseline, Hourly from 0 - 8 hours, 24, 48, and 72 hours, and at 7 days
  Patient self-assessment of pain levels using Visual Analogue Scale
Pulmonary artery pressure assessment | Baseline, Pre-infusion, 1 hour post-infusion
  Trans-thoracic Echocardiography (TTE)

CONTACTS AND LOCATIONS:
Overall Officials: Tania Small, MD, Study Director — Sangart, Inc.
Locations (5):
- Hôpital Henri Mondor, Créteil, France
- Sickle Cell Unit, University of West Indies, Kingston, Jamaica
- Rafic Hariri University Hospital, Beirut, Lebanon
- United Kingdom (2):
  - Guy's Hospital, London
  - King's College London, London

REFERENCES:
- See also: Sangart, Inc. (Home page) — http://www.sangart.com